CLINICAL TRIAL: NCT00167778
Title: Turning Corners: Prosthetic Components and Stability in Amputee Gait
Brief Title: Prosthetic Components and Stability in Amputee Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A3611-R
Record Dates: First submitted 2005-07-01; First posted 2005-09-14 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus; Leg Injuries; Traumatic Amputation
Keywords: Amputation; Amputee; Artificial limbs; Gait; Locomotion; Walking
MeSH Terms: conditions — Diabetes Mellitus; Leg Injuries; Amputation, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Novel prosthetic pylon
  Interventions: Device: Transverse plane rotation adaptor pylon
- Arm 2 (Active Comparator): rigid pylon
  Interventions: Device: Rigid pylon

INTERVENTIONS:
Device: Transverse plane rotation adaptor pylon — Potential future practice
  Arms: Arm 1
Device: Rigid pylon — Current clinical practice
  Arms: Arm 2

SUMMARY:
The biomechanics of changing direction while walking has been largely neglected despite its relevancy to functional mobility. In addition, an increased risk of injury can be associated with turning due to a decrease in stability. The objective of this study is to understand the biomechanics of turning gait in sample populations of intact and trans-tibial amputees and the capacity of prosthetic components to facilitate transverse plane movement. The clinical impact of this investigation is the development of interventions that increase functional mobility, stability and safety while turning.

The researchers propose to investigate three sets of hypotheses. The first set addresses the fundamental biomechanical mechanisms associated with walking along a circular trajectory, how intact subjects differ from amputees, and the effect of a rotation adaptor pylon. The second set of hypotheses addresses dynamic stability and the potential influence of prosthetic interventions. The third set of hypotheses addresses how the rotational properties of the prosthetic pylon can influence comfort and mobility during daily activities.

DETAILED DESCRIPTION:
Most of what is known about how amputees walk and how the properties of prosthetic components affect their gait has been discovered through sagittal plane observations while amputees walk back and forth along a straight line. Abnormal limb loading, thought to be a principal factor in the occurrence of residual limb pain which in turn may cause instability and limit mobility, can certainly occur while walking in a straight line. However, the incidence of abnormal limb loading is likely amplified when performing more complex gait activities, such as turning or avoiding obstacles; activities that are so very common in everyday life.

The specific aims of this investigation are to:

1. discover the biomechanical strategies used and the stability of both intact individuals and trans-tibial amputees walking along a circular trajectory and
2. explore the effects of a prosthetic intervention on turning biomechanics, stability, comfort, and mobility.

We propose to investigate three sets of hypotheses:

The first set of hypotheses addresses the fundamental biomechanical mechanisms associated with walking along a circular trajectory, how intact subjects differ from amputees, and the effect of a rotation adaptor pylon. We will conduct experiments to test three hypotheses related to achieving a change of heading, orientation, and balancing of centripetal forces necessary to walk along a circular trajectory.

The second set of hypotheses seeks to identify whether trans-tibial amputees with a rigid pylon are more unstable during a turning task than non-amputees and whether or not the rotation adaptors enhance stability. We will conduct experiments to calculate an index of dynamic stability that measures the rate at which a person can respond to a perturbation and return to a stable gait pattern.

The third set of hypotheses addresses how the rotational properties of the prosthetic pylon can influence comfort and mobility during daily activities. To measure comfort and mobility, we will solicit questionnaire responses and step count measures from amputees after a one-month period of wearing a rigid pylon and after a one-month period of wearing a transverse plane rotation adaptor (within-subject comparison). In addition to these field measurements, we will also compare the distance traveled during a six-minute walk. Patient opinions about their prosthesis and mobility measures over long periods of time can play a significant role in prosthesis evaluation.

For veteran amputees who experience discomfort and increased risk for residual limb skin problems, it seems reasonable to suppose that these problems might occur when walking along a curved trajectory rather than just a straight line. The joint forces and moments of turning may differ significantly from those exhibited while walking in a straight line. The proposed research will create a new knowledge base with which to understand prosthetic intervention effectiveness. The immediate clinical impact for the trans-tibial amputee is the determination if transverse plane rotational adapter pylons can improve their comfort, mobility, and stability.

ELIGIBILITY:
Inclusion Criteria:

* Amputee Subjects:

  * be a unilateral trans-tibial amputee between the ages of 18 and 70,
  * weigh 220 pounds or less,
  * have been fit with a prosthesis and using a prosthesis for at least two years,
  * wear the prosthesis for at least 8 hours per day,
  * walk without crutches or a walker,
  * able to walk outside the home and in the community,
  * have not fallin within the last six months,
* Non-amputee subjects participating in this investigation will meet similar inclusion criteria except for those related to prosthesis use.

Exclusion Criteria:

* Amputee Subjects:

  * amputation due to tumor, have an active tumor, or are undergoing treatment of a tumor,
  * have pain in legs or any condition that interferes with walking.
* Non-amputee subjects participating in this investigation will meet similar exclusion criteria except for those related to cause of amputation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K. Klute, PhD, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was conducted at the VA Puget Sound Health Care System (Seattle VA hospital). Recruitment began on May 18, 2006. The study was closed to enrollment on April 24, 2008.
  Data was not collected on the order in which participants received each study intervention.
Pre-assignment Details: The prostheses used in this study were built and aligned by a certified and licensed prosthetist prior to beginning starting the protocol. 12 individuals provided informed consent. 1 withdrew prior to starting for personal reasons. 1 withdrew due to unrelated back pain after being fit with both study prostheses and starting with the rigid pylon.
Groups:
- Amputee: This is a randomized cross-over study. Each participant wore both study prostheses: (1) a rigid pylon and (2) a transverse plane torsion adapter. The torsion adapter was initially set according to the manufacturer's recommendations based on body mass and activity level. After one week of acclimation, additional stiffness adjustments were made based on participant feedback. This process continued until the perceived stiffness was optimized. All participants were able to find a comfortable fit either on the first or second visit. Subjects were then randomized, provided with one of two study prostheses, and asked to wear it for 3 weeks. Data was then collected during lab visit 1, and following 1 more week, additional data was collected during lab visit 2. Subjects were then provided with the second study prosthesis and asked to wear it for 3 weeks. Data was then collected during lab visit 3, and following 1 more week, additional data was collected during lab visit 4.
Period: Overall Study
Arm/Group | Amputee
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Amputee: Lower limb amputees who wore both rigid and torsion adapter pylons in random order and completed the study protocol.
Arm/Group | Amputee
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Amputation Etiology [Number; unit: participants]
  Trauma | 5
  Diabetic/Dysvascular | 4
  Tumor | 1
Torsion adapter stiffness [Mean (Standard Deviation); unit: units on a scale] — Settings on the torsion adapter ranged from -5 to 5 in integer increments, where 5 was the stiffest possible setting.
  units on a scale | 4 (2)
Weight [Mean (Standard Deviation); unit: kg] | 88 (11)
Height [Mean (Standard Deviation); unit: m] | 1.79 (.08)

OUTCOME MEASURES:

1. Primary Outcome: Local Dynamic Stability (Hip During Straight Walking)
Description: Maximum finite-time Lyapunov exponents were used to estimate the local dynamic stability of the amputee's sagittal plane hip, knee and ankle angles for their prosthetic limb with and without the torsion adapter while walking straight, while turning with the prosthesis on the inside of the turn, and while turning with the prosthesis on the outside of the turn. Maximum finite-time Lyapunov exponents measure the rate of kinematic separation of a gait cycle trajectory perturbed by naturally occurring disturbances and neuromuscular control errors. A positive exponent indicates divergence of a system, with increasing values indicating a les stable system.
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Groups:
- Rigid Pylon: A rigid pylon is a non-flexible prosthetic component that connects the prosthetic socket to the prosthetic foot.
- Torsion Adapter Pylon: A torsion adapter pylon is a prosthetic component that connects the prosthetic socket to the prosthetic foot and includes a device that allows transverse plane rotation at the socket-pylon interface.
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | .74 (.12) | .74 (.13)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.99, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

2. Primary Outcome: Local Dynamic Stability (Knee During Straight Walking)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | 1.00 (.21) | 1.16 (.30)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

3. Primary Outcome: Local Dynamic Stability (Ankle During Straight Walking)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | .81 (.23) | .96 (.28)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

4. Primary Outcome: Local Dynamic Stability (Hip During Turning With the Prosthesis on the Inside of the Turn)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | .85 (.11) | .83 (.14)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.7, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

5. Primary Outcome: Local Dynamic Stability (Knee During Turning With the Prosthesis on the Inside of the Turn)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | 1.20 (.30) | 1.20 (.25)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.99, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

6. Primary Outcome: Local Dynamic Stability (Ankle During Turning With the Prosthesis on the Inside of the Turn)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | .96 (.22) | .87 (.27)

7. Primary Outcome: Local Dynamic Stability (Hip During Turning With the Prosthesis on the Outside of the Turn)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | .75 (.10) | .74 (.11)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.8, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

8. Primary Outcome: Local Dynamic Stability (Knee During Turning With the Prosthesis on the Outside of the Turn)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | 1.16 (.18) | 1.12 (.29)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.7, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

9. Primary Outcome: Local Dynamic Stability (Ankle During Turning With the Prosthesis on the Outside of the Turn)
Description: as for outcome 1
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
dimensionless | .84 (.33) | .96 (.21)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = .4, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05

10. Secondary Outcome: Peak External Rotation Moment of the Outside Hip While Turning
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: N*mm/kg
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
N*mm/kg | -70 (54) | -88 (45)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.15, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05. Values of p>0.15 were considered not significant (NS) statistically; The effect of study prosthesis was analyzed using repeated measures one-way analyses of variance

11. Secondary Outcome: Peak External Rotation Moment of the Outside Knee While Turning
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: N*mm/kg
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
N*mm/kg | -7 (21) | -15 (15)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.15, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05. Values of p>0.15 were considered not significant (NS) statistically; The effect of study prosthesis was analyzed using repeated measures one-way analyses of variance

12. Secondary Outcome: Peak External Rotation Moment of the Outside Ankle While Turning
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: N*mm/kg
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
N*mm/kg | -28 (31) | -42 (33)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.15, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05. Values of p>0.15 were considered not significant (NS) statistically; The effect of study prosthesis was analyzed using repeated measures one-way analyses of variance

13. Secondary Outcome: Peak External Rotation Moment of the Inside Hip While Turning
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: N*mm/kg
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
N*mm/kg | -54 (47) | -57 (45)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.15, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05. Values of p>0.15 were considered not significant (NS) statistically; The effect of study prosthesis was analyzed using repeated measures one-way analyses of variance

14. Secondary Outcome: Peak External Rotation Moment of the Inside Knee While Turning
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: N*mm/kg
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
N*mm/kg | -26 (27) | -24 (15)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.15, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05. Values of p>0.15 were considered not significant (NS) statistically; The effect of study prosthesis was analyzed using repeated measures one-way analyses of variance

15. Secondary Outcome: Peak External Rotation Moment of the Inside Ankle While Turning
Time Frame: Measurements were taken after wearing the study prostheses for three weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Deviation); unit: N*mm/kg
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
N*mm/kg | -36 (48) | -25 (16)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p > 0.15, Mixed Models Analysis — Statistical significance was set a-prior at p<0.05. Values of p>0.15 were considered not significant (NS) statistically; The effect of study prosthesis was analyzed using repeated measures one-way analyses of variance

16. Secondary Outcome: Activity Level
Description: Average number of steps per day over a 1 week period ending in the fourth week of each study prosthesis (Rigid and Torsion adapter)
Time Frame: One week
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Error); unit: Steps/day
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
Steps/day | 6269 (1080) | 6728 (1121)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.05; Wilcoon paired signed rank test for the differences between Rigid and Torsion Adapter pylons

17. Secondary Outcome: Six-minute Walk Distance
Description: Participants are asked to walk alone as far as possible without running for six minutes. This test is performed indoors along a long, flat straight hallway of approximately 30 meters in length with two orange cones marking the 180 degree turnaround points at each end of the corridor. Approximately 40 straight steps were taken for every four turning steps.
Time Frame: Six minutes after wearing the study prostheses for four weeks.
Population: Each participant wore both study prostheses.
Measure: Mean (Standard Error); unit: m
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 10 | 10
m | 463 (24) | 464 (26)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.05; Wilcoxon paired signed rank test for the differences between Rigid and Torsion Adapter pylons

18. Secondary Outcome: Residual Limb Pain at Present?
Description: The residual limb pain grade scores ranged from 0 "No Pain/ Interference" to 10 "Severe Pain/Interference."
Time Frame: Measurements were taken after wearing the study prostheses for four weeks
Population: 10 participants wore both study prostheses but only 7 participants presented with pain.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 7 | 7
units on a scale | 2.0 (0.7) | 1.6 (0.7)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.1; Wilcoxon paired signed rank test for the differences between the Rigid and Torsion Adapter pylons

19. Secondary Outcome: Average Residual Limb Pain?
Description: The residual limb pain grade scores ranged from 0 "No Pain/ Interference" to 10 "Severe Pain/Interference."
Time Frame: Measurements were taken after wearing the study prostheses for four weeks.
Population: 10 participants wore both study prostheses but only 7 participants presented with pain.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 7 | 7
units on a scale | 2.9 (0.5) | 2.3 (0.6)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.1; Wilcoxon paired signed rank test for the differences between the Rigid and Torsion Adapter pylons

20. Secondary Outcome: Worst Residual Limb Pain?
Description: The residual limb pain grade scores ranged from 0 "No Pain/ Interference" to 10 "Severe Pain/Interference."
Time Frame: Measurements were taken after wearing the study prostheses for four weeks.
Population: 10 participants wore both study prostheses but only 7 participants presented with pain.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 7 | 7
units on a scale | 4.7 (1.0) | 3.6 (0.7)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.1; Wilcoxon paired signed rank test for the differences between the Rigid and Torsion Adapter pylons

21. Secondary Outcome: Least Residual Limb Pain?
Description: The residual limb pain grade scores ranged from 0 "No Pain/ Interference" to 10 "Severe Pain/Interference."
Time Frame: Measurements were taken after wearing the study prostheses for four weeks.
Population: 10 participants wore both study prostheses but only 7 participants presented with pain.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 7 | 7
units on a scale | 1.9 (0.6) | 1.6 (0.6)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.1; Wilcoxon paired signed rank test for the differences between the Rigid and Torsion Adapter pylons

22. Secondary Outcome: Pain Interference With Activities?
Description: The residual limb pain grade scores ranged from 0 "No Pain/ Interference" to 10 "Severe Pain/Interference."
Time Frame: Measurements were taken after wearing the study prostheses for four weeks.
Population: 10 participants wore both study prostheses but only 7 participants presented with pain.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 7 | 7
units on a scale | 3.4 (0.8) | 1.6 (0.6)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.057, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.1; Wilcoxon paired signed rank test for the differences between the Rigid and Torsion Adapter pylons

23. Secondary Outcome: How Bothersome Was Your Pain?
Description: The residual limb pain grade scores ranged from 0 "No Pain/ Interference" to 10 "Severe Pain/Interference."
Time Frame: Measurements were taken after wearing the study prostheses for four weeks.
Population: 10 participants wore both study prostheses but only 7 participants presented with pain.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Rigid Pylon | Torsion Adapter Pylon
Number analyzed (Participants) | 7 | 7
units on a scale | 3.1 (1.1) | 2.9 (1.1)
Statistical Analysis 1: Comparison: Rigid Pylon vs Torsion Adapter Pylon; Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney) — Statistical significance was set a-prior at p<0.1; Wilcoxon paired signed rank test for the differences between the Rigid and Torsion Adapter pylons

ADVERSE EVENTS:
Arm/Group | Amputee
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Our sample population consisted of community ambulators whose results may not generalize to all lower limb amputees.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes